CLINICAL TRIAL: NCT07134140
Title: Effects of Omega-3 Fatty Acid Supplementation on Muscle Performance, Neuromuscular Function, and Inflammation at Rest and Following Eccentric Exercise.
Brief Title: Omega-3 Fatty Acids in Muscle Function and Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Responsible Party: Principal Investigator, Dr. Anastasios Theodorou, Associate Professor, European University Cyprus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EUC omega-3
Record Dates: First submitted 2025-08-10; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: omega-3; eccentric exercise; muscle function
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega-3 (Experimental): Participants in this group will take 3 g of fish oil [(NOW, Ultra Omega-3 Fish Oil, (NOW, Bloomingdale, IL, USA)] for 12 weeks.
  Interventions: Dietary Supplement: Omega-3
- Placebo (Placebo Comparator): Participants in this group will take 3 g of olive oil for 12 weeks.
  Interventions: Dietary Supplement: Placebo comparator

INTERVENTIONS:
Dietary Supplement: Omega-3 — Participants will take three capsules per day (a total of 1,500 mg EPA and 750 mg DHA). They will take 1 g with each main meal (breakfast, lunch, and dinner).
  Arms: Omega-3
Dietary Supplement: Placebo comparator — Participants will take 3 g of olive oil. They will take 1 g with each main meal (breakfast, lunch, and dinner).
  Arms: Placebo

SUMMARY:
This study aims to investigate the effects of omega-3 fatty acid supplementation on muscle performance, neuromuscular function, inflammation, and oxidative stress at rest and after eccentric exercise. The findings may provide insights into the role of omega-3 fatty acids in muscle function, physiology, and metabolism following muscle-damaging exercise. Additionally, the effects of omega-3 fatty acids on cardiovascular health will be investigated.

DETAILED DESCRIPTION:
The study is a double-blind, randomized controlled trial. Two parallel groups of 16 healthy males and females each (sex counterbalanced, 20-45 years) will randomly take 3 g of fish oil [1500 mg EPA (eicosapentaenoic acid) + 750 mg DHA (docosahexaenoic acid), Now Foods, USA] or a placebo (3 g of olive oil) for 12 weeks. Before taking the supplement, participants will perform a unilateral isokinetic eccentric exercise session of maximal voluntary intensity (10 repetitions x 10 sets of knee extensions at a speed of 60 degrees per second). Dominant and non-dominant legs will be allocated equally and randomly across participants. Physiological assessments and blood samples will be collected immediately before exercise and 2 and 4 days after eccentric exercise (bout 1). Then, participants will start the supplementation for 12 weeks. At the end of the supplementation period, participants will perform the same eccentric exercise protocol (bout 2) with their opposite leg. The same assessments and blood sampling will be conducted at the same time points (i.e., immediately before and 2 and 4 days after eccentric exercise).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) within the normal range (18.5-25 kg/m²).
* Healthy individuals without severe medical conditions (e.g., diabetes, coronary artery disease, hypertension, neuromuscular disorders).
* No musculoskeletal injury in the lower limbs (e.g., bone fracture, tendon rupture, grade III muscle strain) within the last 6 months before enrollment.
* Negative responses to all questions on the PAR-Q questionnaire indicating no contraindications to participating in exercise testing.
* Mentally capable of providing informed consent.

Exclusion Criteria:

* Use of any pharmaceutical medications (e.g., statins, aspirin, ibuprofen).
* Use of dietary supplements (e.g., protein, vitamins) within the last 3 months before enrollment.
* Participation in a structured training program involving more than three training sessions per week during the study period.
* Following a special diet (e.g., intermittent fasting, ketogenic diet, vegetarian diet).
* Allergy or intolerance to fish oil or olive oil.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | Changes in muscle strength after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Muscle strength of the knee extensors will be measured using an isokinetic dynamometer during maximal voluntary contractions. The unit of measure is Newton-meters (Nm).
Maximal Oxygen Uptake (VO₂ max) | Changes in VO₂ max after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  VO₂ max will be assessed during a graded exercise test on a cycle ergometer. The measure unit is milliliters per kilogram of body mass per minute (ml/kg/min).
Muscle Fatigue Index (MFI) | Changes in MFI after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  MFI will be calculated as the percentage decline (%) in peak torque across a series of repeated maximal contractions of the knee extensor muscles on an isokinetic dynamometer.
Muscle Oxygenation | Changes in muscle oxygenation after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Muscle oxygenation will be measured in the vastus lateralis using near-infrared spectroscopy (NIRS). Parameters include oxyhemoglobin (O₂Hb), deoxyhemoglobin (HHb), and total hemoglobin levels, which will be expressed in arbitrary units (AU).
Creatine Kinase | Change in creatine kinase activity after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Creatine kinase activity will be measured in International Units (IU) via the enzymatic colorimetric method in fasting plasma samples.
Range of Motion (ROM) | Change in ROM after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  ROM of the knee joint will be measured in degrees (°) using an isokinetic dynamometer, with full extension defined as 0° and flexion recorded up to 120°.
Muscle Thickness | Change in muscle thickness after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Muscle thickness of the vastus lateralis will be measured using B-mode ultrasound with a linear probe, in millimeters (mm).
Echo Intensity | Change in echo intensity after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Echo intensity of the vastus lateralis will be assessed using B-mode ultrasound with a linear probe and quantified from grayscale image analysis, expressed in arbitrary units (0-255).
Blood Lipids Profile | Change in blood lipids from baseline (immediately before supplementation) to 12 weeks after the supplementation period.
  Fasting blood samples will be collected and analyzed to assess the participant's lipid profile, including: Total Cholesterol (TC). Expressed in mg/dL. Low-Density Lipoprotein Cholesterol (LDL-C). Expressed in mg/dL. High-Density Lipoprotein Cholesterol (HDL-C). Expressed in mg/dL. Triglycerides (TG). Expressed in mg/dL. Blood will be drawn after a minimum of 8-12 hours of fasting. Lipid concentrations will be determined using standard enzymatic colorimetric methods on an automated clinical chemistry analyzer.

SECONDARY OUTCOMES:
Omega-3 Index | Change in omega-3 index in red blood cells from baseline (immediately before supplementation) to 12 weeks after the supplementation period.
  The Omega-3 Index will be assessed as a biomarker of long-chain omega-3 fatty acid status. It is defined as the combined percentage (%) of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in red blood cell (RBC) membranes, expressed as a proportion of total identified fatty acids.
  Blood samples will be collected following an overnight fast, and red blood cells will be isolated for fatty acid analysis. EPA and DHA levels will be quantified via gas chromatography, and the Omega-3 Index will be reported as a percentage (%).
Rate of Force Development (RFD). | Change in RFD after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  RFD will be calculated as the slope of the torque-time curve during the early phase of voluntary contraction. It will be measured in Newton-meters per second (Nm/s).
Electromechanical Delay (EMD) | Change in EMD after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  EMD will be defined as the time lag between the onset of electrical activity (via surface EMG) and the onset of force production, measured in milliseconds (ms).
Force Matching Error (FME) | Change in FME after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  FME will be assessed during a submaximal isometric contraction using an isokinetic dynamometer and expressed as the percentage difference between the target and produced force (%).
Joint Position Sense (JPS) | Change in JPS after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  JPS will be evaluated as the absolute angular difference between a target knee joint angle and the participant's reproduced angle, measured in degrees (°) using an isokinetic dynamometer.
Delayed Onset Muscle Soreness (DOMS). | Change in DOMS after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  DOMS will be assessed using a 1-10 visual analog scale (VAS), where 1 indicates no pain and 10 indicates extreme pain.
Countermovement Jump (CMJ) | Change in CMJ after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  CMJ will be measured in centimeters (CM) using a force plate.
Contact Time | Change in contact time after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Duration of foot contact with the force plate during landing, expressed in milliseconds (ms).
Stability Index | Change in stability index after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  The stability index will be assessed from the center of pressure displacement using a force platform and expressed in millimeters (mm).
F2-Isoprostanes | Change in F2-Isoprostanes after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  F2-Isoprostanes will be quantified as a marker of lipid peroxidation using ELISA and expressed in picograms per milliliter (pg/mL).
Glutathione | Change in glutathione after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Glutathione will be measured as an indicator of endogenous antioxidant capacity using a colorimetric assay and expressed in micromoles per gram of hemoglobin (μmol/g Hb).
Protein carbonyls | Change in protein carbonyls after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Protein carbonyls will be measured as a marker of oxidative protein damage using a spectrophotometric assay and expressed in nanomoles per gram of hemoglobin (nmol/g Hb).
Interleukin-6 (IL-6) | Change in IL-6 after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  IL-6 will be measured as a marker of inflammation using ELISA and expressed in picograms per milliliter (pg/mL).
Tumor Necrosis Factor-alpha (TNF-α) | Change in TNF-α after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  TNF-α will be measured as a marker of inflammation using ELISA and expressed in picograms per milliliter (pg/mL).
Pennation Angle | Change in pennation angle after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  The pennation angle of the vastus lateralis will be measured under resting conditions using longitudinal B-mode ultrasound imaging and expressed in degrees (°).
Fascicle Length | Change in fascile length after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Fascicle length of the vastus lateralis will be determined under resting condition from B-mode ultrasound images, either measured directly from visible fascicles or estimated using trigonometric calculations, and expressed in millimeters
Muscle Stiffness | Change in muscle stifness after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Muscle stiffness, reflecting the resistance of the muscle to an external force, will be measured and expressed in newtons per meter (N/m) using the Myoton Pro device.
Muscle Tone | Change in muscle tone after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Muscle tone will be assessed using the Myoton Pro device, representing the natural oscillation frequency of the muscle at rest, and expressed in hertz (Hz).
Mechanical Stress Relaxation Time | Change in mechanical stress relaxation time after the first bout (week 0) and the second bout of exercise (week 12) from baseline (immediately before each bout) and at day 2 and day 4 after each exercise bout.
  Mechanical stress relaxation time will be assessed using the Myoton Pro device, representing the time required for the muscle to return to its original shape after a mechanical impulse, and expressed in milliseconds (ms).
Central and Peripheral Blood Pressure | Change in blood pressure from baseline (immediately before supplementation) to 12 weeks after the supplementation period.
  Central and peripheral systolic and diastolic blood pressure will be measured using the SphygmoCor system and expressed in millimeters of mercury (mmHg).
Arterial stiffness | Change in arterial stiffness from baseline (immediately before supplementation) to 12 weeks after the supplementation period.
  Arterial stiffness will be assessed using the SphygmoCor system by measuring carotid-femoral pulse wave velocity (PWV), expressed in meters per second (m/s).

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios A Theodorou, Dr., Study Chair — European University Cyprus
Locations (1):
- European University Cyprus, Nicosia, Engomi, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results will be shared as supplementary files in accordance with the policies of each journal. Data sharing may vary across publications based on journal-specific requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified dataset and supporting documentation will be made available beginning after the publication of the primary study results in a peer-reviewed journal, or within 24 months of final study completion (whichever occurs first). Data will remain accessible for 10 years thereafter.
Access Criteria: De-identified individual participant data and supporting documentation (study protocol, statistical analysis plan, dataset) will be available to qualified researchers conducting methodologically sound proposals. Access will be granted after approval of a data access request and completion of a data use agreement. Data will be accessible through a secure institutional repository.